CLINICAL TRIAL: NCT02618941
Title: Phase IB Follow-up, Controlled, Parallel Group, Single-center Study to Assess a Second Boost Immunization With AFFITOPE® PD01A With Regard to Safety/Tolerability, Immunological and Clinical Activity in Patients Who Have Participated in the AFF008 Program
Brief Title: Follow-up Study to Assess a Second Boost Immunization With AFFITOPE® PD01A With Regard to Safety and Clinical Activity (AFF008AA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFFiRiS 008AA; 2015-004854-16 (EudraCT Number)
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AFFITOPE® PD01A + Adjuvant (Experimental): one injection of 75µg AFFITOPE® PD01A/adjuvanted
  Interventions: Biological: AFFITOPE® PD01A
- Control (No Intervention): Untreated control group

INTERVENTIONS:
Biological: AFFITOPE® PD01A — s.c. injection
  Arms: AFFITOPE® PD01A + Adjuvant

SUMMARY:
This is a follow-up study to assess safety and clinical activity of continued AFFITOPE® PD01A vaccinations in patients with Parkinson's disease. Patients, who have already participated in the AFF008 program will be involved and will receive a second boost immunization with AFFITOPE® PD01A. One study site in Vienna (Austria) will be involved.

In addition, up to 6 patients will be offered participation within an untreated control Group.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in AFF008, AFF008E and AFF008A
* Written informed consent signed and dated by the patient and, preferentially, the caregiver
* In the investigator's opinion, does not have visual or auditory impairments that would reduce the patients' ability to complete study questionnaires or be unable to receive instructions for These
* Female patients of childbearing potential are eligible if they use a medically accepted contraceptive method
* All changes in conventional PD therapies must be available to the sponsor; in particular pharmacologic symptomatic PD medication allowing transformation to a Levodopa standard dose
* A potential participant should be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history (except PD therapies, these will be recorded separately) for at least 30 days prior to Visit 1 if considered relevant by the investigator

Exclusion Criteria:

* Women of childbearing potential without birth control or pregnant women
* Participation in another clinical trial within 3 months before Visit 1 (except AFF008A)
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial
* Autoimmune disease or allergy to components of the vaccine
* History of cancer (Exceptions: non-melanoma skin cancer, intraepithelial cervical neoplasia)
* Active infectious disease (e.g., Hepatitis B, C)
* Immunodeficiency
* Significant systemic illness
* Alcoholism or substance abuse
* Prior and/or current treatment with experimental immunotherapeutics including IVIG with the exception of AFFITOPE® PD01A, with immune modulating drugs or treatment with deep brain stimulation
* Venous status rendering it impossible to place an i.v. access

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of any Serious Adverse Events (SAE) that are related to the study drug | 12 months
Number of patients who withdraw due to Adverse Events (AEs) | 12 months
  The withdrawal criteria (continuation decision) in regards to the number of patients who withdraw due to AEs as well as the reason for withdrawal will be evaluated.
Occurrence of any Grade 3 or higher AEs related to the study drug within 4 weeks after vaccination | 12 months

SECONDARY OUTCOMES:
Immunological activity of AFFITOPE® vaccine PD01A | 12 months
  Titer of vaccination induced antibodies directed towards vaccine components and the target (native aSyn) assessed by ELISA (or equivalent method)

OTHER OUTCOMES:
MDS-UPDRS Ia, II, III | 12 months
  Change in motor/non-motor symptoms over time
PDQ39 | 12 months
  Change in non-motor PD symptoms over time
PD NMS | 12 months
  Change in non-motor PD symptoms over time
Cognitive scales | 12 months
  Change in non-motor PD symptoms over time

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Volc, Prim. Dr., Principal Investigator — Studienzentrum der PROSENEX, AmbulatoriumsbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt
Locations (1):
- Studienzentrum der PROSENEX, AmbulatoriumsbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt, Vienna, Austria

REFERENCES:
- [Derived] McFarthing K, Simuni T. Clinical Trial Highlights: Targetting Alpha-Synuclein. J Parkinsons Dis. 2019;9(1):5-16. doi: 10.3233/JPD-189004. No abstract available. PMID 30741694